CLINICAL TRIAL: NCT04184947
Title: Cardiovascular Outcomes of Type 2 Diabetic Patients Treated With SGLT-2 Inhibitors Versus GLP-1 Receptor Agonists in Real-life. An Observational Study Using Clinical-administrative Data
Brief Title: Cardiovascular Outcomes SGLT-2 Inhibitors Versus GLP-1 Receptor Agonists
Status: Completed | Type: Observational
Sponsor: University of Padova (Other)
Responsible Party: Sponsor
Other Study IDs: DIMEDDEI3
Record Dates: First submitted 2019-12-01; First posted 2019-12-04 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SGLT2i: Patients who received new prescription of a SGLT-2 inhibitor
  Interventions: Drug: SGLT2 inhibitor
- GLP-1RA: Patients who received new prescription of a GLP-1 receptor agonist
  Interventions: Drug: GLP-1 receptor agonist

INTERVENTIONS:
Drug: SGLT2 inhibitor — New prescription of a SGLT-2 inhibitor (dapagliflozin, empagliflozin or canagliflozin) at any dosage during routine clinical practice
  Groups: SGLT2i
Drug: GLP-1 receptor agonist — New prescription of a GLP-1 receptor agonisty (exenatide, liraglutide, lixisenatide, dulaglutide) at any dosage during routine clinical practice
  Groups: GLP-1RA

SUMMARY:
Patients with type 2 diabetes (T2D) suffer from an excess risk of adverse cardiovascular events. Recently, two classes of glucose lowering agents, namely SGLT-2 inhibitors (SGLT2i) and GLP-1 receptor agonists (GLP-1RA), have proved superior to placebo in protecting T2D patients from cardiovascular events in dedicated trials. Patient populations in such trials were mainly composed of T2D individuals with established cardiovascular disease (CVD) or at very high risk for CVD. In addition, no clinical trial has so far compared cardiovascular outcomes of T2D associated with SGLT2i versus GLP-1RA. In addition, whether different results would incur in patients at lower CVD risk is unclear. On this basis, we designed this retrospective real-world study to compare cardiovascular outcomes of patients newly treated with SGLT2i versus GLP-1RA in routine clinical practice

ELIGIBILITY:
Inclusion Criteria:

* Italian citizens, residing in the Region
* Registered as beneficiaries for at least one year between January 1st, 2012 and September 30th, 2018
* Diagnosis of type 2 diabetes
* Newly initiating SGLT-2 inhibitors or GLP-1 receptor agonists
* Being treated with glucose lowering medications before (at least one prescription of an antidiabetic agent in ATC class A10B prior to the index date)
* Time between the index date and the last SGLT2 inhibitors or GLP-1 receptor agonists prescription shorter than 8 months,
* Follow-up time or time-to-endpoint of at least three months

Exclusion Criteria:

* Patients who started SGLT2i or GLP-1RA before 2014
* Patients with an insufficient exposure time
* Patients with an incident event within three months after the index date.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Type 2 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
3 point major adverse cardiovascular events (4P-MACE) | 3-26 months after index date
  First occurrence of myocardial infarction, stroke, or death

SECONDARY OUTCOMES:
Hospitalization for cardiovascular causes | 3-26 months after index date
  First hospitalization for any cardiovascular cause
Death | 3-26 months after index date
  All-cause death
Myocardial infarction | 3-26 months after index date
  Myocardial infarction
Heart failure | 3-26 months after index date
  Hospitalization for heart failure
Stroke | 3-26 months after index date
  Stroke or transient ischemic attack
Revascularization | 3-26 months after index date
  Any arterial site revascularization (surgical or endovascular)

OTHER OUTCOMES:
Occurrence of adverse events | 3-26 months after index date
  Occurrence of: amputation, Fournier's gangrene, bone fracture, diabetic ketoacidosis, infections, pancreatitis, pancreatic cancer, acute kidney injury

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Metabolic Diseases, University Hospital of Padova, Padua, Italy

IPD SHARING:
Plan to Share IPD: No
Data cannot be shared

REFERENCES:
- [Derived] Longato E, Di Camillo B, Sparacino G, Gubian L, Avogaro A, Fadini GP. Cardiovascular outcomes of type 2 diabetic patients treated with SGLT-2 inhibitors versus GLP-1 receptor agonists in real-life. BMJ Open Diabetes Res Care. 2020 Jun;8(1):e001451. doi: 10.1136/bmjdrc-2020-001451. PMID 32591373